CLINICAL TRIAL: NCT03253380
Title: Targets Of Early Rehabilitation Program In Critically Ill Chronic Obstructed Airway Disease Patients
Brief Title: Early Rehabilitation Program In Critically Ill Chronic Obstructed Airway Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hend mohammed sayed mohammed (Other)
Responsible Party: Sponsor-Investigator, Hend mohammed sayed mohammed, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17100100
Record Dates: First submitted 2017-08-10; First posted 2017-08-17 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- early rehabilitation program on mechanical ventilated COPD pat (Experimental): compare the effect of early rehabilitation program on mechanical ventilated COPD patient in RICU to those using current standard care as regarding (morbidity and thirty day mortality ,diaphragm function and weaning outcomes, disease exacerbation , Duration spent on machin , Length of ICU stay.
  Interventions: Other: Early Rehabilitation Program In Critically Ill Chronic Obstructed Airway Disease patients

INTERVENTIONS:
Other: Early Rehabilitation Program In Critically Ill Chronic Obstructed Airway Disease patients — Early rehabilitation of MV patients in the respiratory ICU

SUMMARY:
this study aim to compare the effect of early rehabilitation program on mechanical ventilated COPD patient in Respiratory ICU to those using current standard care as regarding :

* morbidity and thirty day mortality
* diaphragm function and weaning outcomes.
* disease exacerbation
* Duration spent on ventilator.
* Length of ICU stay

DETAILED DESCRIPTION:
Mechanical ventilation (MV) in intensive care units (ICUs) essential in the management of respiratory failure, can result in respiratory dysfunction and inspiratory muscle weakness. Like any other striated muscle, respiratory muscle mass is affected by contractile inactivity. In fact, the respiratory muscles appear more sensitive to the effects of disuse compared with other striated muscles .

In humans, relatively brief periods of diaphragm disuse (<3 days) due to controlled mechanical ventilation are associated with diaphragm muscle fiber atrophy , force-generating capacity of the diaphragm was reduced by ±32 % after 5-6 days of controlled mechanical ventilation in intensive care unit (ICU) patients.

the degree of weakness is correlated with the duration of ventilation. One case-control study demonstrated that MV results in increased proteolysis and atrophy in the diaphragm muscle, while other skeletal muscles are spared .Respiratory muscle weakness is associated with adverse clinical outcomes, including difficult weaning from mechanical ventilation, increased mortality, and increased risk of ICU/hospital readmission .

Inspiratory muscle training (IMT) has been used in patients with chronic lung disease for many years, resulting in not just increased inspiratory muscle strength but also increased inspiratory muscle endurance, reduced dyspnoea and increased exercise tolerance and quality of life.

Early rehabilitation of MV patients in the ICU has been claimed not only to be safe but to reduce ICU length of stay, decrease time spent on MV, and improve outcomes after discharge

The primary aim of this study is To compare the effect of early rehabilitation program on mechanical ventilated COPD (chronic obstructive pulmonary disease ) patient in RICU (respiratory intensive care unit )to those using current standard care as regarding :

* morbidity and thirty day mortality
* diaphragm function and weaning outcomes.
* disease exacerbation
* Duration spent on machine .
* Length of ICU stay.

The Secondary aim is to Establish the HRQoL and physical function critical care survivors up to six months after ICU discharge

All patients will be subjected to the following:

1. Initial assessment: (general and local chest examination, laboratory investigations in the form of: arterial blood gases serum electrolytes, liver and kidney functions, blood glucose, complete blood picture, chest radiography (Antro-posterior view),ECG)
2. standard medical treatment in the form of: (antibiotics bronchodilators corticosteroids expectorants, prophylactic anticoagulant) participants will be randomly assigned to receive either standard care plus comprehensive pulmonary rehabilitation or standard care alone

The patients will be categorized into 2 groups according to simplicity of weaning:

Group I: ) participants will be receive standard care plus comprehensive pulmonary rehabilitation Group II: ) participants will be receive current standard care .

Pulmonary rehabilitation intervention:

sedation hold then assessment of the patient using the Richmond Agitation-Sedation Scale(RASS). to achieve a sedation level of 'easily aroused and cooperative'(RASS of -1, 0 or +1). If the sedation hold is successful, the participant will be screened for safety to start of rehabilitation.

Participants meeting any of the following criteria will fail the safety screen:

* mean arterial pressure (MAP) <65 mm Hg;
* heart rate <40 or>130 bpm
* respiratory rate <5 or >40 breaths/min;
* marked ventilator asynchrony;
* oxygen saturation <88%
* active gastrointestinal bleeding;
* acute myocardial ischemia;
* agitation requiring increased sedatives

The participant must be able to obey at least three of the following commands:

1. opening eyes in response to voice;
2. using eyes to follow investigator on request;
3. squeezing hand on request and
4. protruding tongue on request. If the participant can follow at least three of these commands and has a RASS of -1, 0 or +1, they will be achieved 'wakefulness', and pulmonary rehabilitation will be started.

Upper and lower limb exercise activity events: sit on the edge of hospital bed without back support, sit in a chair after transfer from the hospital bed, and ambulate with or without assistance using a walker and/or support from the RICU staff.

Respiratory muscle exercise:

Usual physiotherapy care typically involves - Percussion

* deep breathing exercises
* manual hyperinflation ( delivery of a slow inspiration, a 2-3 s inspiratory hold, and a fast uninterrupted expiratory flow that mimics a forced expiration).
* secretion clearance techniques,
* In mechanical ventilated patient Respiratory muscle training will be based on increasing the trigger sensitivity gradually in order to I increase muscle endurance. The trigger sensitivity was adjusted to 20% of the first recorded MIP at the start of training (In the first session), inspiratory muscle training (IMT) was limited to 5 min; afterwards the duration was increased by 5 min at every session until it reached 30 min . . If a patient tolerated 30 min of IMT, The next session would be performed with increasing trigger sensitivity by 10% of the initial MIP .Patients who could not tolerate IMT with 20% of MIP for 5 min were trained with 10% of MIP IMT sessions stopped after 5 days and trial of weaning was done

The training session was interrupted when the treating therapist observed any of the following:

1. respiratory rate greater than 35 breaths/min or 50% higher than at the start of the session.
2. oxygenated haemoglobin saturation less than 90%; systolic pressure greater than 180 mmHg or less than 80 mmHg.
3. heart rate more than 140beats/min or 20% higher than at the start of the session.
4. paradoxical breathing; agitation; depression haemoptysis; arrhythmia or sweating

   Pulmonary rehabilitation program (include patients on non invasive ventilation and patient weaned from mechanical ventiltion

   ) Duration period: at least 6 days

   Breathing Exercises:

   • Have the patient assume a comfortable, relaxed position and loosen restrictive clothing. Initially, a semi-Fowler's position with the head and trunk elevated approximately 45, is desirable. By supporting the head and trunk, flexing the hips and knees, and supporting the legs with a pillow, the abdominal muscles remain relaxed.
   * Other positions, such as supine, sitting, or standing, may be used initially or as the patient progresses during treatment.
   * Pay attention to relaxation of the sternocleidomastoids, upper trapezius, and levator scapulae muscles . Never allow a patient to force or prolonged expiration. Expiration should be relaxed or lightly controlled Do not allow the patient to initiate inspiration with the accessory muscles and the upper chest Allow the patient to perform deep breathing for only three or four inspirations and expirations at a time to avoid hyperventilation

   GLOSSOPHARYNGEAL BREATHING It is a technique that is performed by using the muscles of mouth, cheeks, lips, tongue, soft palate, larynx and pharynx to piston boluses of air into the lungs.

   Diaphragmatic breathing:

   Diaphragmatic breathing enhance diaphragmatic descent during inspiration and diaphragmatic ascent during expiration 5 minutes about 3 times per day.

   Pursed Lip Breathing:

   Have the patient breathe in slowly and deeply through the nose and then breathe out gently through lightly pursed lips as if blowing on and bending the flame of a candle but not blowing it out Teaching an Effective Cough Have the patient assume a relaxed, comfortable position for deep breathing and coughing.

   Sitting or leaning forward usually is the best position for coughing. The patient's neck should be slightly flexed to make coughing more comfortable. Teach the patient controlled diaphragmatic breathing, emphasizing deep inspirations Have the patient place the hands on the abdomen and make three huffs with expiration When the patient has put these actions together, instruct the patient to take a deep but relaxed inspiration, followed by a sharp double cough

   • Manual-Assisted Cough • If a patient has abdominal weakness (e.g., as the result of a mid-thoracic or cervical spinal cord injury), manual pressure on the abdominal area assists in developing greater intra-abdominal pressure for a more forceful cough.

   Sandbag Breathing:

   In the last 2 days of the rehab program. Done three times daily use light weighted sandbag, about 1-2 kilograms The sandbag is put on the patient's upper abdomen just below the xiphoid process and the patient is asked to practice diaphragmatic breathing for 2 minutes followed by a minute off weight breathing. Repeat the previous step once again.
   * Research outcome measures:

     a. Primary (main): effect of pulmonary rehabilitation in comparison to standard care group by the following:

1-the duration of the period of weaning from mechanical ventilation, duration of ICU stay and duration of hospital stay.

2-RICU morbidity and thirty day mortality

3-1st readmission in ER, ward, ICU during 1st 6 months of discharge. 4-.Respiratory muscle strength and function by I) Maximal inspiratory pressure (MIP) will be measured to evaluate global respiratory muscle strength High values for MIP exclude clinically significant weakness.

II) Chest Ultrasonography for assessment of diaphragm function using these views:

1-. subcostal view:

* reduced caudal movement of the diaphragm during unassisted breathing is (weakness)
* paradoxal movement (diaphragm paralysis). 2 Mid axillary view Diaphragm atrophy will be assessed by measuring diaphragm thickness in the mid axillary line at the level of the diaphragm dome and its thickening fraction during inspiration to asses contractile activity 5-Physical and mental health as measured by the Short Form 36 Health Survey (SF-36)

ELIGIBILITY:
Inclusion Criteria:

* All COPD patients admitted to ICU are aged more than 18 years are haemodynamically stable and requiring minimal ventilatory support (ie positive end expiratory pressure (PEEP) less than or equal100.

Exclusion Criteria:

* medically unstable (eg, new cardiac arrhythmia , heamodynamic unstable)
* experiencing significant pain that interferes with breathing capacities, fractured ribs
* have major disorders which affect the central nervous system resulting in permanent weakness that is not responsive to exercise training
* COPD patient with neuromuscular disease or overlap with OSA (obstructive sleep apnea).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Measure thirty day mortality rate among COPD patients who was subjected to early rehabilitation program during mechanical ventilation in RICU and those using current standard care | 2 years
  measure the percentage of patients who die within 30 days after mechanical ventilation
Measure disease exacerbation among COPD patients who was subjected to early rehabilitation program during mechanical ventilation in RICU and those using current standard care | 2 years
  measure number of exacerbations in COPD patients during six months after weaning from mechanical ventilation
Measure duration spent on ventilator among COPD patients who was subjected to early rehabilitation program during mechanical ventilation in RICU and those using current standard care | 2 years
  measure duration of mechanical ventilation
Measure duration of ICU stay among COPD patients who was subjected to early rehabilitation program during mechanical ventilation in RICU and those using current standard care | 2 years
  measure duration of ICU stay